CLINICAL TRIAL: NCT06122441
Title: RE-inventing Strategies for Healthy Ageing; Recommendations and Tools (RESTART) - a Randomized Controlled Trial Testing a Complex Lifestyle Intervention in Older Adults at Increased Risk for Cardiometabolic Disease
Brief Title: RE-inventing Strategies for Healthy Ageing; Recommendations and Tools
Acronym: RESTART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Research Council of Norway (Other); Novo Nordisk A/S (Industry); Tromso Municipality (Unknown); University Hospital of North Norway (Other); University of Oslo (Other); Molde University College (Other); National Association for Heart and Lung Diseases, Tromso, Norway (Unknown); Norwegian Trekking Association (Unknown); KRAFT Sports Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/584841(REK)
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Lifestyle, Healthy; Muscle Weakness; Abdominal Obesity; Cardiometabolic Syndrome; Self Efficacy; Diet, Healthy
Keywords: Complex lifestyle intervention; Older adults; Cardiometabolic risk factors; Cardiorespiratory fitness; Muscle strength; Physical activity; Abdominal obesity; Acceptance and commitment therapy; Health-related quality of life; Cognitive function
MeSH Terms: conditions — Muscle Weakness; Obesity, Abdominal; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: RESTART is designed as a two-arm, single blind, parallel group RCT, with a 1:1 allocation ratio into either intervention or active control group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group assignment from baseline to primary endpoint assessment. It is not possible to blind the participants or intervention staff due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex lifestyle intervention (Experimental): Receives a complex lifestyle intervention, a wrist-worn activity tracker, and access to national recommendations on physical activity.
  Interventions: Behavioral: Complex lifestyle intervention; Behavioral: Physical activity monitoring and recommendations
- Active control (Active Comparator): Receives a wrist-worn activity tracker and access to national recommendations on physical activity.
  Interventions: Behavioral: Physical activity monitoring and recommendations

INTERVENTIONS:
Behavioral: Complex lifestyle intervention — The complex lifestyle intervention comprise high-intensity aerobic and strength exercise, behavioral counselling based on Acceptance and Commitment Theory (ACT), and dietary counselling based on Norwegian nutritional guidelines. The different intervention elements are introduced step-wise to reduce initial overload. Participants are progressively transitioned over to the Tromsø municipality and local NGO's, who delivers activities harmonized with the intervention elements. Participants are at this stage also supported by an eTool which digitally reinforces the intervention through web-based information and videos.
  Arms: Complex lifestyle intervention
Behavioral: Physical activity monitoring and recommendations — Wrist-worn activity trackers that are worn throughout the trial, which monitors steps, activity intensity and energy expenditure. Access to Norwegian physical activity guidelines via the Directorate of Health.

SUMMARY:
The goal of the RESTART RCT is to examine whether a complex lifestyle intervention, coordinated with municipal and non-government organizations (NGO), can establish and preserve improvements in risk factors and functional capacity among older adults at high risk of cardiometabolic disease. The main objectives to investigate are whether a complex lifestyle intervention, compared to an active control group, will at 24 months have:

1. Produced a clinically relevant increase in cardiorespiratory fitness (primary endpoint)
2. Increased muscle strength, physical activity and reduced adiposity
3. Improved body composition, health-related quality of life and cognitive function

All participants (Control and Intervention Groups) are provided with wrist-worn activity trackers at baseline and access to national recommendations on physical activity. The intervention group additionally advances through a comprehensive lifestyle program including high-intensity aerobic and strength exercise, dietary and behavioral counselling. Intervention participants are gradually transitioned into exercise activities organized by Tromsø Municipaity and local NGO:s. Testing of outcomes are performed at baseline, 6, 12 and 24 months. Primary endpoint (VO2max) is assessed at 24 months.

DETAILED DESCRIPTION:
The proportion of older individuals worldwide is growing, posing a significant challenge to western societies. To address the health challenges of the aging population, primary prevention efforts should focus on various lifestyle factors simultaneously. However, many interventions fail to maintain improved lifestyle habits among participants, highlighting the need for novel and complex approaches to ensure healthy aging among older adults.

The RESTART randomized controlled trial aims to investigate whether participants undergoing a complex lifestyle intervention improve their cardiorespiratory fitness, muscle strength, physical activity, adiposity and body composition, quality of life and cognitive function at 24 months, compared to active controls.

The study and data collection will occur in Tromsø, Norway (pop. 77,000). Participants will receive the intervention at a local community exercise center near the University of Tromsø campus area. Testing of physical performance will take place at the UiT Faculty of Health Sciences research laboratory for sports, physical activity, and public health. The Clinical Trial Unit (CTU) at the local university hospital will additionally oversee clinical examinations, collection of questionnaire data, and blood sampling.

At baseline, both the Control and Intervention Groups are given wrist-worn activity trackers and access to national physical activity recommendations. The Intervention Group also undergoes a comprehensive lifestyle program that includes high-intensity aerobic and strength exercises, as well as dietary and behavioral counseling. The Intervention Group is gradually introduced to exercise activities organized by Tromsø Municipality and local NGOs. Outcome testing is conducted at baseline, 6, 12, and 24 months, with the primary endpoint (VO2max) assessed at 24 months.

Intervention participants will be divided into 4 groups of 12-15 participants each and perform high-intensity training to target the cardiovascular system and skeletal muscle force-generating capacity. For 12 months, the intervention group performs supervised indoor cycling or outdoor hill interval training twice a week at a relatively high intensity (≥85% of maximal heart rate during 4x4 minutes) separated by active rest periods at approximately 70% of maximal heart rate. Immediately after the aerobic exercise, participants perform strength training (3 sets of 5 repetitions) involving leg-press, lateral pull-down, and chest press exercises, with an intensity corresponding to ≥80% of their maximal strength. From months 6-12, one of the two weekly exercise sessions will be led by the Healthy Life Center (HLC; "Frisklivssentralen"), enabling a transition to supervised exercise via the Tromsø municipality primary health care. Between month 12-18, the HLC continue to supervise the participants during one weekly exercise sessions, while they are additionally introduced to exercise activities arranged by local NGO:s.

From month 3 to 12, participants will receive behavioral counseling based on the Acceptance and Commitment Therapy (ACT) approach during six 2-hour group sessions. The individual approach aims to enhance participants' capacity to manage challenging cognitive and emotional experiences, foster psychological flexibility and distress tolerance skills, and promote the development of self-efficacy and new behavior patterns that align with their life values.

From month 6 to 12, the intervention group will receive four dietary counseling sessions based on Norwegian nutritional guidelines. Two individual sessions will involve food diaries, while two group sessions with a partner will focus on basic nutritional information and practical food preparation. The objective is to promote a healthy, sustainable, and personalized diet while promoting increased protein intake, reducing the consumption of high-energy-dense foods and drinks with low nutritional value.

Beginning from month 12 and onwards throughout the trial, the intervention group will be granted access to the Re-start eTool (https://re-start.no/), which is specifically tailored to older adults. The eTool offers concise and easy-to-understand articles, videos, and self-assessment tools that promote physical activity, healthy dietary habits, and behavioral strategies from the complex intervention. The Re-start eTool aims to provide support and reminders to participants as they gradually transition to independently maintaining the achieved lifestyle habits and physical capacity levels.

Throughout the study period, the intervention instructors and assessors monitor potential adverse events during the exercise and testing phases, and all adverse events are reported to the study coordinator. Measures to mitigate adverse events include: 1) insurance of participants via The Norwegian System of Patient Injury Compensation; 2) involving a MD with sports medicine specialization to ensure treatment of potential injuries; 3) pilot study experiences show that short-term alternative exercises are effective in managing exercise-induced pain and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75 years
* BMI ≥ 30 kg/m2
* Elevated CVD-risk (Score 8/12 on the NORRISK 2 model)
* Sedentary lifestyle (Score "1" on the Saltin-Grimby Physical Activity Level Scale)

Exclusion Criteria:

* Presence of dementia diagnosis
* Self-reported previous myocardial infarction or stroke, and/or self-reported established cardiovascular disease by presence of coronary stent
* Heart failure with ejection fraction <50%
* Electrocardiogram ECG presenting with atrioventricular block grade 2 type 2 or grade 3, or previous myocardial infarction.
* Uncontrolled hypertension (systolic blood pressure≥180 mmHg and/or diastolic blood pressure≥110 mmHg unless cleared by a nephrologist)
* Chronic obstructive pulmonary disease grade 3 or 4
* Thyroid dysfunction (thyroxine <7 pmol/L and thyroid-stimulating hormone >10 mIU/L, and/or thyroxine >25 pmol/L and thyroid-stimulating hormone <0.2 mIU/L)
* Liver dysfunction (alanine aminotransferase >210 µmol/L for men, >135 µmol/L for women, and/or aspartate aminotransferase >135 µmol/L for men, >105 µmol/L for women, and/or alkaline phosphatase >345 µmol/L)
* Kidney dysfunction (creatinine >220 µmol/L), in addition to prognosis of CKD by GFR and Albuminuria KDIGO 2012 algorithm
* Severe anemia (hemoglobin <10g/dL for men, <8g/dL for women)
* Uncontrolled diabetes (glycated hemoglobin ≥86 mmol/mol)
* Severe hearing problems
* Severe mobility limitations (unable to get up from a sitting or lying position, unable to maintain a crouched position, unable to raise arms above shoulder or head height)
* No possession of a smartphone
* No access to the Norwegian national identification service (BankID)
* Unable to follow the trial regimen for 24 months

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in VO2max at month 24 | Baseline and month 24
  Assessed as ml/kg/min during an incremental test-to-exhaustion where the participant walks or runs on a motorized treadmill.
Change from baseline in VO2max at month 12 | Baseline and month 12
  Assessed as ml/kg/min during an incremental test-to-exhaustion where the participant walks or runs on a motorized treadmill.
Change from baseline in VO2max at month 6 | Baseline and month 6
  Assessed as ml/kg/min during an incremental test-to-exhaustion where the participant walks or runs on a motorized treadmill.

SECONDARY OUTCOMES:
Change from baseline in muscle strength at month 24 | Baseline and month 24
  Assessed as the highest kg achieved during a 1-repetition maximum test in leg-press and chest-press apparatuses.
Change from baseline in muscle strength at month 12 | Baseline and month 12
  Assessed as the highest kg achieved during a 1-repetition maximum test in leg-press and chest-press apparatuses.
Change from baseline in muscle strength at month 6 | Baseline and month 6
  Assessed as the highest kg achieved during a 1-repetition maximum test in leg-press and chest-press apparatuses.
Change from baseline in muscle power at month 24 | Baseline and month 24
  Assessed as power (W; force x speed of contraction) during leg-press exercise with pre-defined weight ascertained during baseline measurements
Change from baseline in muscle power at month 12 | Baseline and month 12
  Assessed as power (W; force x speed of contraction) during leg-press exercise with pre-defined weight ascertained during baseline measurements
Change from baseline in muscle power at month 6 | Baseline and month 6
  Assessed as power (W; force x speed of contraction) during leg-press exercise with pre-defined weight ascertained during baseline measurements
Change from baseline in waist circumference at month 24 | Baseline and month 24
  Assessed in centimeters at the umbilical level (between crista iliaca and the lower rib) using a measurement tape.
Change from baseline in waist circumference at month 12 | Baseline and month 12
  Assessed in centimeters at the umbilical level (between crista iliaca and the lower rib) using a measurement tape.
Change from baseline in waist circumference at month 6 | Baseline and month 6
  Assessed in centimeters at the umbilical level (between crista iliaca and the lower rib) using a measurement tape.
Change from baseline in body weight at month 24 | Baseline and month 24
  Assessed in kilograms using a SECA personal weight. Participants are measured without outdoor clothing and shoes.
Change from baseline in body weight at month 12 | Baseline and month 12
  Assessed in kilograms using a SECA personal weight. Participants are measured without outdoor clothing and shoes.
Change from baseline in body weight at month 6 | Baseline and month 6
  Assessed in kilograms using a SECA personal weight. Participants are measured without outdoor clothing and shoes.
Change from baseline in minutes in moderate-to-vigorous physical activity per day at month 24 | Baseline and month 24
  Assessed as minutes in light, moderate and vigorous intensity, using triaxial accelerometers worn at the hip for 7 days.
Change from baseline in minutes in moderate-to-vigorous physical activity per day at month 12 | Baseline and month 12
  Assessed as minutes in light, moderate and vigorous intensity, using triaxial accelerometers worn at the hip for 7 days.
Change from baseline in minutes in moderate-to-vigorous physical activity per day at month 6 | Baseline and month 6
  Assessed as minutes in light, moderate and vigorous intensity, using triaxial accelerometers worn at the hip for 7 days.
Daily physical activity pattern | 24 months
  Asessed using wrist-worn smartwatches that are worn by the participants continously and measures steps, activity intensity and energy expenditure

OTHER OUTCOMES:
Change from baseline in relative body composition at month 24 | Baseline and month 24
  Assessed as percentage fat and lean mass in relation to total body mass using Dual-Energy X-ray Absorptiometry
Change from baseline in relative body composition at month 12 | Baseline and month 12
  Assessed as percentage fat and lean mass in relation to total body mass using Dual-Energy X-ray Absorptiometry
Change from baseline in absolute body composition at month 24 | Baseline and month 24
  Assessed as fat/lean/bone mass in grams using Dual-Energy X-ray Absorptiometry
Change from baseline in absolute body composition at month 12 | Baseline and month 12
  Assessed as fat/lean/bone mass in grams using Dual-Energy X-ray Absorptiometry
Change from baseline in health-related quality of life at month 24 | Baseline and month 24
  Assessed with a 5-point likert scale in 5 different dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) using the EQ-5D-5L instrument
Change from baseline in health-related quality of life at month 12 | Baseline and month 12
  Assessed with a 5-point likert scale in 5 different dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) using the EQ-5D-5L instrument
Change from baseline in cognitive function using the Digit Symbol Substitution Test at month 24 | Baseline and month 24
  Assessed as the number of symbols correctly matched with numbers within the allowed time
Change from baseline in cognitive function using the Digit Symbol Substitution Test at month 12 | Baseline and month 12
  Assessed as the number of symbols correctly matched with numbers within the allowed time
Change from baseline in forced expiratory volume (FEV1) at month 24 | Baseline and month 24
  Assessed as litres/sec using the Micro 1 Spirometer with participants exhaling maximally for six seconds during three attempts with 30 seconds of rest in between.
Change from baseline in forced vital capacity (FVC) at month 24 | Baseline and month 24
  Assessed as litres using the Micro 1 Spirometer with participants exhaling maximally for six seconds during three attempts with 30 seconds of rest in between.
Change from baseline in peak expiratory flow (PEF) at month 24 | Baseline and month 24
  Assessed as litres/min using the Micro 1 Spirometer with participants exhaling maximally for six seconds during three attempts with 30 seconds of rest in between.
Change from baseline in resting heart rate at month 24 | Baseline and month 24
  Assessed as beats per minute three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in resting heart rate at month 12 | Baseline and month 12
  Assessed as beats per minute three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in resting heart rate at month 6 | Baseline and month 6
  Assessed as beats per minute three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in systolic and diastolic blood pressure at month 24 | Baseline and month 24
  Assessed as mmHg three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in systolic and diastolic blood pressure at month 12 | Baseline and month 12
  Assessed as mmHg three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in systolic and diastolic blood pressure at month 6 | Baseline and month 6
  Assessed as mmHg three times in 1-minute intervals after an initial 2-minute rest
Change from baseline in hand-held dynamometer-derived maximal handgrip strength at month 24 | Baseline and month 24
  Assessed in kg and performed according to the Southampton protocol
Change from baseline in hand-held dynamometer-derived maximal handgrip strength at month 12 | Baseline and month 12
  Assessed in kg and performed according to the Southampton protocol
Change from baseline in 5-repetition chair stand test performance at month 24 | Baseline and month 24
  Assessed as time (s) to complete 5 consecutive chair rises, using the 5-repetition chair stand test according to the Short Physical Performance Battery protocol
Change from baseline in 5-repetition chair stand test performance at month 12 | Baseline and month 12
  Assessed as time (s) to complete 5 consecutive chair rises, using the 5-repetition chair stand test according to the Short Physical Performance Battery protocol
Change from baseline in satisfaction with life at month 24 | Baseline and month 24
  Assessed with a 7-point likert scale using the 5-item Satisfaction With Life Scale (SWLS)
Change from baseline in satisfaction with life at month 12 | Baseline and month 12
  Assessed with a 7-point likert scale using the 5-item Satisfaction With Life Scale (SWLS)
Change from baseline in mental distress on the 10-item Hopkins Symptom Checklist (HSCL-5) at month 24 | Baseline and month 24
  Assessed with a 5-point likert scale using the 10-item Hopkins Symptom Checklist (HSCL-5)
Change from baseline in mental distress on the 10-item Hopkins Symptom Checklist (HSCL-5) at month 12 | Baseline and month 12
  Assessed with a 5-point likert scale using the 10-item Hopkins Symptom Checklist (HSCL-5)
Change from baseline in physical activity discomfort and acceptance on the 10-item Physical Activity Acceptance Questionnaire (PAAQ) at month 24 | Baseline and month 24
  Assessed with a 7-point likert scale using the 10-item Physical Activity Acceptance Questionnaire (PAAQ)
Change from baseline in physical activity discomfort and acceptance on the 10-item Physical Activity Acceptance Questionnaire (PAAQ) at month 12 | Baseline and month 12
  Assessed with a 7-point likert scale using the 10-item Physical Activity Acceptance Questionnaire (PAAQ)
Change from baseline in physical activity enjoyment on the 4-item Physical Activity Enjoyment Scale Short Form (PACES-S) at month 24 | Baseline and month 24
  Assessed with a 4-point likert scale using the 4-item Physical Activity Enjoyment Scale Short Form (PACES-S)
Change from baseline in physical activity enjoyment on the 4-item Physical Activity Enjoyment Scale Short Form (PACES-S) at month 12 | Baseline and month 12
  Assessed with a 4-point likert scale using the 4-item Physical Activity Enjoyment Scale Short Form (PACES-S)
Change from baseline in emotional eating on the 3-item Emotional Eating Subscale from the Three-Factor Eating Questionnaire (TFEQ) at month 24 | Baseline and month 24
  Assessed with a 4-point likert scale using the 3-item Emotional Eating Subscale from the Three-Factor Eating Questionnaire (TFEQ)
Change from baseline in emotional eating on the 3-item Emotional Eating Subscale from the Three-Factor Eating Questionnaire (TFEQ) at month 12 | Baseline and month 12
  Assessed with a 4-point likert scale using the 3-item Emotional Eating Subscale from the Three-Factor Eating Questionnaire (TFEQ)
Change from baseline in binge eating episodes on the Eating Disorder Examination (EDE) questionnaire at month 24 | Baseline and month 24
  Assessed with a 7-point likert scale using the item on binge eating episodes from the Eating Disorder Examination (EDE) questionnaire
Change from baseline in binge eating episodes on the Eating Disorder Examination (EDE) questionnaire at month 12 | Baseline and month 12
  Assessed with a 7-point likert scale using the item on binge eating episodes from the Eating Disorder Examination (EDE) questionnaire
Change from baseline in intuitive eating on the 6-item Reliance on Internal Hunger and Satiety Cues Subscale from the Intuitive Eating Scale (IES) at month 24 | Baseline and month 24
  Assessed with a 5-point likert scale using the 6-item Reliance on Internal Hunger and Satiety Cues Subscale from the Intuitive Eating Scale (IES)
Change from baseline in intuitive eating on the 6-item Reliance on Internal Hunger and Satiety Cues Subscale from the Intuitive Eating Scale (IES) at month 12 | Baseline and month 12
  Assessed with a 5-point likert scale using the 6-item Reliance on Internal Hunger and Satiety Cues Subscale from the Intuitive Eating Scale (IES)
Change from baseline in self-efficacy on the 10-item General Self-Efficacy Scale (GSE) at month 24 | Baseline and month 24
  Assessed with a 4-point likert scale using the 10-item General Self-Efficacy Scale (GSE)
Change from baseline in self-efficacy on the 10-item General Self-Efficacy Scale (GSE) at month 12 | Baseline and month 12
  Assessed with a 4-point likert scale using the 10-item General Self-Efficacy Scale (GSE)
Change from baseline in self-compassion on the 6-item Self-Compassion Scale at month 24 | Baseline and month 24
  Assessed with a 5-point likert scale using the 6-item Self-Compassion Scale
Change from baseline in self-compassion on the 6-item Self-Compassion Scale at month 12 | Baseline and month 12
  Assessed with a 5-point likert scale using the 6-item Self-Compassion Scale
Change from baseline in self-reported education status at month 24 | Baseline and month 24
  Assessed using 4 alternatives (from elementary school to college/university) using the education status question from a standardized comprehensive questionnaire from the 7th data collection wave of the Tromsø Study (2015-2016)
Change from baseline in self-reported household income at month 24 | Baseline and month 24
  Assessed with a 8-point likert scale using the household income question from a standardized comprehensive questionnaire from the 7th data collection wave of the Tromsø Study (2015-2016)
Change from baseline in self-reported occupation status at month 24 | Baseline and month 24
  Assessed with 9 nominal alternatives without intrinsic order using the occupation status question from a standardized comprehensive questionnaire from the 7th data collection wave of the Tromsø Study (2015-2016)
Change from baseline in self-reported occupation status at month 12 | Baseline and month 12
  Assessed with 9 nominal alternatives without intrinsic order using the occupation status question from a standardized comprehensive questionnaire from the 7th data collection wave of the Tromsø Study (2015-2016)
Change from baseline in self-reported occupation status at month 6 | Baseline and month 6
  Assessed with 9 nominal alternatives without intrinsic order using the occupation status question from a standardized comprehensive questionnaire from the 7th data collection wave of the Tromsø Study (2015-2016)
Change from baseline in self-reported ideal weight at month 24 | Baseline and month 24
  Assessed using a 5-item questionnaire on ideal weight combining 2 dichotomous (yes/no) scales and 3 continuous scales. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported ideal weight at month 12 | Baseline and month 12
  Assessed using a 5-item questionnaire on ideal weight combining 2 dichotomous (yes/no) scales and 3 continuous scales. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported chronic disease at month 24 | Baseline and month 24
  Assessed using a 11-item questionnaire with each item including a 3-point ordinal scale response option (no, yes-previously, yes-now). This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported chronic disease at month 12 | Baseline and month 12
  Assessed using a 11-item questionnaire with each item including a 3-point ordinal scale response option (no, yes-previously, yes-now). This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported symptoms and complaints at month 24 | Baseline and month 24
  Assessed using a 10-item questionnaire including 8 items with dichotomous response alternatives and 6 items with ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported symptoms and complaints at month 12 | Baseline and month 12
  Assessed using a 10-item questionnaire including 7 items with dichotomous response alternatives and 3 items with ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported medicine use at month 24 | Baseline and month 24
  Assessed using a 9-item questionnaire including 8 items with ordinal scale response alternatives and 1 item with free text response alternative to list currently used medicine. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported medicine use at month 12 | Baseline and month 12
  Assessed using a 9-item questionnaire including 8 items with ordinal scale response alternatives and 1 item with free text response alternative to list currently used medicine. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported medicine use at month 6 | Baseline and month 6
  Assessed using a 9-item questionnaire including 8 items with ordinal scale response alternatives and 1 item with free text response alternative to list currently used medicine. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported social network at month 24 | Baseline and month 24
  Assessed using a 4-item questionnaire including 3 items with nominal scale response alternatives and 1 item with ordinal scale response alternative. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported social network at month 12 | Baseline and month 12
  Assessed using a 4-item questionnaire including 3 items with nominal scale response alternatives and 1 item with ordinal scale response alternative. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported tobacco use at month 24 | Baseline and month 24
  Assessed using a 2-item questionnaire including ordinal scale response alternatives (never, yes-previously, yes-now). This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported tobacco use at month 12 | Baseline and month 12
  Assessed using a 2-item questionnaire including ordinal scale response alternatives (never, yes-previously, yes-now). This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported alcohol use at month 24 | Baseline and month 24
  Assessed using a 3-item questionnaire with ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported alcohol use at month 12 | Baseline and month 12
  Assessed using a 3-item questionnaire with ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-rated health at month 24 | Baseline and month 24
  Assessed using a 2-item questionnaire with 5-point ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-rated health at month 12 | Baseline and month 12
  Assessed using a 2-item questionnaire with 5-point ordinal scale response alternatives. This questionnaire was developed as part of the comprehensive standardized questionnaire used in the 7th data collection wave of the Tromsø Study (2015-2016).
Change from baseline in self-reported leisure time physical activity level at month 24 | Baseline and month 24
  Assessed using the 4-item Saltin-Grimby Physical Activity Level Scale
Change from baseline in self-reported leisure time physical activity level at month 12 | Baseline and month 12
  Assessed using the 4-item Saltin-Grimby Physical Activity Level Scale
Change from baseline in self-reported diet using the NORKOST Food Frequency Questionnaire at month 24 | Baseline and month 24
  Assessed using the Norwegian NORKOST Food Frequency Questionnaire including 274 items on various food groups and specific foods
Change from baseline in self-reported diet using the NORKOST Food Frequency Questionnaire at month 12 | Baseline and month 12
  Assessed using the Norwegian NORKOST Food Frequency Questionnaire including 274 items on various food groups and specific foods
Change from baseline in hemoglobin (Hb) and glycated hemoglobin (HbA1C) at month 24 | Baseline and month 24
  Assessed as % using non-fasted blood samples analysed with high-performance liquid chromatography
Change from baseline in hemoglobin (Hb) and glycated hemoglobin (HbA1C) at month 12 | Baseline and month 12
  Assessed as % using non-fasted blood samples analysed with high-performance liquid chromatography
Change from baseline in hemoglobin (Hb) and glycated hemoglobin (HbA1C) at month 6 | Baseline and month 6
  Assessed as % using non-fasted blood samples analysed with high-performance liquid chromatography
Change from baseline in blood lipids (total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides) at month 24 | Baseline and month 24
  Assessed as mmol/l using non-fasted blood samples analysed with colorimetric (Homogen, or homogen enzymatic) methods
Change from baseline in blood lipids (total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides) at month 12 | Baseline and month 12
  Assessed as mmol/l using non-fasted blood samples analysed with colorimetric (Homogen, or homogen enzymatic) methods
Change from baseline in blood lipids (total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides) at month 6 | Baseline and month 6
  Assessed as mmol/l using non-fasted blood samples analysed with colorimetric (Homogen, or homogen enzymatic) methods
Change from baseline in renal function markers (cystatin C, creatinine) at month 24 | Baseline and month 24
  Collected as non-fasting venous blood samples using standard methods
Change from baseline in renal function markers (cystatin C, creatinine) at month 12 | Baseline and month 12
  Collected as non-fasting venous blood samples using standard methods
Change from baseline in renal function markers (cystatin C, creatinine) at month 6 | Baseline and month 6
  Collected as non-fasting venous blood samples using standard methodsdescribed
Baseline levels of markers of thyroid function (thyroxin, thyroid-stimulating hormone) | Baseline
  Collected as non-fasting venous blood samples using standard methods. Used primarily as a potential exclusion criteria.
Change from baseline in liver enzymes (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase) at month 24 | Baseline and month 24
  Collected as non-fasting venous blood samples using standard methods
Change from baseline in liver enzymes (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase) at month 12 | Baseline and month 12
  Collected as non-fasting venous blood samples using standard methods
Change from baseline in phosphatidylethanol at month 24 | Baseline and month 24
  Collected as a non-fasting venous blood sample using standard methods in order to monitor alcohol consumption
Change from baseline in phosphatidylethanol at month 12 | Baseline and month 12
  Collected as a non-fasting venous blood sample using standard methods in order to monitor alcohol consumption
Change from baseline in testosterone at month 24 | Baseline and month 24
  Collected as a non-fasting venous blood sample using standard methods
Change from baseline in testosterone at month 12 | Baseline and month 12
  Collected as a non-fasting venous blood sample using standard methods
Change from baseline in C-reactive protein at month 24 | Baseline and month 24
  Collected as a non-fasting venous blood sample using standard methods
Change from baseline in C-reactive protein at month 12 | Baseline and month 12
  Collected as a non-fasting venous blood sample using standard methods
Change from baseline in albumin-creatinine ratio at month 24 | Baseline and month 24
  Collected as a morning urine sample using standard methods
Change from baseline in albumin-creatinine ratio at month 12 | Baseline and month 12
  Collected as a morning urine sample using standard methods
Change from baseline in albumin-creatinine ratio at month 6 | Baseline and month 6
  Collected as a morning urine sample using standard methods
Change from baseline in ECG PQ-interval at month 24 | Baseline and month 24
  Assessed in milliseconds using a 12-point electrocardiogram (ECG) to evaluate the time interval from the beginning of the P wave to the beginning of the QRS complex, to establish atrioventricular block (grade 1-3)
Change from baseline in ECG P-wave at month 24 | Baseline and month 24
  Assessed in milliseconds using a 12-point electrocardiogram (ECG) to evaluate the atrial depolarization, and used to determine cardiac rhythm disturbance (atrial fibrillation)
Change from baseline in ECG QRS-complex at month 24 | Baseline and month 24
  Assessed in milliseconds using a 12-point electrocardiogram (ECG) to evaluate the characterization of the QRS-complex to determine ventricular tachycardia
Change from baseline in ECG T-wave at month 24 | Baseline and month 24
  Assessed in millivolts using a 12-point electrocardiogram (ECG) to determine T-wave inversion in V3-6 (negative from baseline)
Participants' experiences of receiving a complex lifestyle intervention | 24 months
  Assessed using qualitative semi-structured interviews to provide a more comprehensive understanding of participants' experiences and motivation during the trial, and to find potential important determinants of lifestyle change. Qualitative data will be structured with the QRS NVivo software, and analyzed with content- or thematic analyses.
Assessment of the cost-effectiveness of receiving the intervention versus not receiving the intervention, over a 24-month period | 24 months
  Data on resource use will be collected during the trial to facilitate health economic evaluation of the personalized lifestyle program. The trial has already mentioned collection of data on health-related quality of life (EQ-5D-5L) that allows us to calculate Quality-Adjusted Life Years, and to subsequently calculate cost-effectiveness (Cost per Quality-Adjusted Life Years).
Number of participants with CVD events (myocardial infarction, stroke), diabetes and premature deaths | 60 months
  Assessed using linkage to the Norwegian Patient Registry and the Norwegian Cause of Death Registry.
Number of participants with intervention-related adverse events | 24 months
  Monitored consequently by intervention and outcome assessment personell

CONTACTS AND LOCATIONS:
Overall Officials: Sameline Grimsgaard, PhD, Principal Investigator — UiT The Arctic University of Norway; Jonas Johansson, PhD, Study Director — UiT The Arctic University of Norway; Trygve Deraas, PhD, Study Director — UiT The Arctic University of Norway; Camilla Flåten, MSc, Study Director — UiT The Arctic University of Norway; André Henriksen, PhD, Study Director — UiT The Arctic University of Norway; Laila Hopstock, PhD, Study Director — UiT The Arctic University of Norway
Locations (1):
- UiT The Arctic University of Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators will have access to the final, complete trial dataset. Other investigators can apply to the steering committee for data and may receive access to data with variables specific to the research question of interest.
Supporting Information: Study Protocol, ICF
Time Frame: From January 2027 until December 2030. A possible extension to 2035 is planned to be applied for from the regional ethics committee
Access Criteria: Anonymous datasets are shared directly via study coordinator. Unidentified datasets (containing potential reverse-identifiable data) are accessed via the Norwegian Services for Sensitive Data server.

REFERENCES:
- [Derived] Johansson J, Deraas TS, Hopstock LA, Henriksen A, Grimsgaard S. Improving and preserving cardiorespiratory fitness, muscle strength and adiposity through a complex lifestyle intervention in community-dwelling older adults with elevated cardiometabolic risk: study protocol for the RESTART randomised controlled trial. BMJ Open. 2025 Apr 19;15(4):e095810. doi: 10.1136/bmjopen-2024-095810. PMID 40254301
- See also: Project webpage (only currently available in Norwegian) — https://uit.no/project/restart

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT06122441/Prot_SAP_001.pdf